CLINICAL TRIAL: NCT04899479
Title: Peri-tREatment of SGLT-2 Inhibitor on Myocardial Infarct Size and Remodeling Index Measured by Cardiac maGnetic rEsonance Imaging in Patients With Acute Myocardial Infarction and High Risk of Heart Failure Undergoing Percutaneous Coronary Intervention
Brief Title: Peri-treatment of SGLT-2 Inhibitor on Myocardial Infarct Size and Remodeling Index in Patients With Acute Myocardial Infarction and High Risk of Heart Failure Undergoing Percutaneous Coronary Intervention
Acronym: PRESTIGE-AMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Bin Song, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESTIGE-AMI
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Percutaneous Coronary Intervention; Infarct size; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Randomization will be performed 1:1 between SGLT-2 inhibitor and control. Stratification will be done by DM and clinical presentation (STEMI vs. NSTEMI).
Masking Description: This is an open-label study, therefore, no masking will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT-2 inhibitor (Experimental): The SGLT-2 inhibitor group will receive SGLT-2 inhibitor once daily until the end of the study period.
  Interventions: Drug: SGLT2 inhibitor
- Control (Placebo Comparator): The control group will not receive any additional drugs.
  Interventions: Other: Control

INTERVENTIONS:
Drug: SGLT2 inhibitor — In patients with AMI and high risk of heart failure, 1:1 randomization will be performed to either SGLT2 inhibitor or control group.
  Arms: SGLT-2 inhibitor
Other: Control — In patients with AMI and high risk of heart failure, 1:1 randomization will be performed to either SGLT2 inhibitor or control group.
  Arms: Control

SUMMARY:
We aimed to identify whether SGLT-2 inhibitor administration before and after coronary intervention is effective in reducing the size of infarction and myocardial remodeling in patients with acute myocardial infarction (AMI) and high risk of heart failure, and its mechanism. For this reason, we compared cardiac magnetic resonance imaging (CMR) parameters and clinical outcomes between the SGLT-2 inhibitor group and the control group to confirm the efficacy and safety of SGLT-2 inhibitors.

DETAILED DESCRIPTION:
After the introduction of percutaneous coronary intervention (PCI) as a method to normalize blood flow in the treatment of coronary artery disease, not only the technical aspects of coronary intervention but also the devices and medications have been improved over the past 30 years. However, despite these advances, morbidity, and mortality of AMI are still high. In particular, in patients with ST-segment elevation MI (STEMI), the 1-year mortality rate and hospitalization rate due to heart failure are 10%, and 22%, respectively. Accordingly, various efforts are being made to improve the prognosis of AMI and to reduce the infarct size, which is a major prognostic factor. The most effective method for achieving this goal to early and successful revascularization by PCI. However, restoring blood flow, which is a prerequisite for relieving ischemia, can paradoxically cause damage to the myocardium and death of the myocardium by itself. This phenomenon is called myocardial reperfusion injury. Several pharmacological and mechanical treatments targeting this phenomenon have been studied, and the experimental and small-scale clinical trials have been shown to have the effect of reducing infarct size and relieving myocardium.4 However, to date, large-scale clinical trials have not demonstrated clinical benefits.

SGLT-2 inhibitors are developed to lower blood sugar and treat type 2 diabetes mellitus (DM) by inhibiting Sodium glucose co-transporter-2 in proximal renal tubule, releasing glucose into the urine and preventing reabsorption. However, SGLT-2 inhibitors are known to have an effect on lowering cardiovascular events in addition to lowering blood sugar. In three large-scale, multicenter, randomized trials to evaluate the effects of SGLT-2 in type 2 diabetic patients, the combined outcome consisting of cardiac death or readmission due to heart failure was significantly lowered compared to the placebo group. In particular, DECLARE-TIMI 58 trial confirmed that this effect was consistent regardless of the history of atherosclerotic cardiovascular disease or heart failure.8 In addition, DAPA-CKD trial showed that SGLT-2 inhibitor significantly reduced the composite outcome consisting of cardiovascular death or readmission due to heart failure as well as the kidney-related outcome compared to the placebo group in patients with chronic kidney disease regardless of type 2 DM. Similarly, EMPEROR-Reduced and DAPA-HF trials consistently demonstrated that SGLT-2 inhibitor was associated with significantly lower risk of a composite of cardiovascular death or worsening heart failure in patients with heart failure with reduced ejection fraction. Therefore, the current guideline recommended the use of SGLT-2 inhibitor in patients with heart failure with reduced ejection fraction, with a conjunction of goal-directed medical therapy. Nevertheless, the mechanism that can explain this has been extensively investigated, but it is not clear yet. Several potential hypotheses have been proposed as mechanisms such as increased natriuresis, decreased blood pressure, decreased inflammation, and decreased reactive oxidative stress. In this regard, it is anticipated that the use of SGLT-2 inhibitors will benefit even in patients with AMI and high risk of heart failure in both acute and chronic phases.

Therefore, we aimed to identify whether SGLT-2 inhibitor administration before and after coronary intervention is effective in reducing the size of infarction and myocardial remodeling in patients with AMI and high risk of heart failure, and its mechanism. For this reason, we compared CMR parameters and clinical outcomes between the SGLT-2 inhibitor group and the control group to confirm the efficacy and safety of SGLT-2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subject must be at least 18 years of age 2) Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving SGLT-2 inhibitor and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure 3) Diagnosis of Type 1 myocardial infarction (MI) (ST-segment elevation MI [STEMI] or Non-ST-segment elevation MI [NSTEMI]) i) Detection of a rise and/or fall of cardiac troponin values with at least 1 value above the 99th percentile upper reference limit ii) Symptoms or electrocardiographic changes suggesting myocardial ischemia 4) High risk of heart failure (at least one of the two criteria below are met) i) Left ventricular ejection fraction < 50% ii) Symptoms or signs of pulmonary congestion requiring treatment

Exclusion Criteria:

* 1) Target lesion is not suitable for PCI by operator's decision 2) Patients requiring cardiopulmonary resuscitation due to cardiac arrest before randomization 3) Rescue PCI after thrombolysis or facilitated PCI 4) Previous MI 5) Previous history of heart failure 6) Patients who have been taking SGLT-2 inhibitor 7) Patients with glomerular filtration rate < 30ml/min/1.73m2 or on dialysis 8) Type 1 diabetes mellitus (DM) 9) Known hypersensitivity or contraindications to study medications (SGLT-2 inhibitor) 10) Pregnant or lactating women 11) Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial infract size (IS) | at 6-month follow-up
  IS measured using CMR
∆Left ventricular end-systolic volume | Between index hospitalization and 6-month follow-up
  Difference of left ventricular end-systolic volume measured by CMR

SECONDARY OUTCOMES:
Acute kidney injury | Within 3 days after index PCI
  According to KDIGO guideline
Myocardial IS | Within 3 days after index PCI
  IS measured using CMR
Microvascular obstruction (MVO) | Within 3 days after index PCI
  MVO measured using CMR
IS | Within 3 days after index PCI
  measured by peak cardiac enzyme
∆left ventricular end-diastolic volume | Between index hospitalization and 6-month follow-up
  Difference of left ventricular end-diastolic volume measured using CMR
∆left ventricular ejection fraction | Between index hospitalization and 6-month follow-up
  Difference of left ventricular ejection fraction measured using CMR
LV adverse remodeling | Between index hospitalization and 6-month follow-up
  measured by CMR
LV reverse remodeling | Between index hospitalization and 6-month follow-up
  measured by CMR
MVO | at 6-month follow-up
  measured using CMR
Changes of NT-proBNP level | Between index hospitalization and 6-month follow-up
  Difference of NT-proBNP
Estimated glomerular filtration rate | 6 months after index PCI
  Kidney function
Cardiovascular death, myocardial infarction, cerebrovascular events, stent thrombosis, and re-hospitalization due to cardiac cause | 12 months after index PCI
  MACE
Cardiovascular death, or re-hospitalization due to cardiac cause | 12 months after index PCI
  cardiovascular death or re-hospitalization due to cardiac cause
All-cause death | 12 months after index PCI
  All-cause death during follow-up
Cardiovascular death | 12 months after index PCI
  Cardiovascular death during follow-up
MI | 12 months after index PCI
  MI during follow-up
Repeat revascularization | 12 months after index PCI
  Repeat revascularization during follow-up
Re-hospitalization due to heart failure | 12 months after index PCI
  Re-hospitalization due to heart failure during follow-up
Re-hospitalization due to cardiac cause | 12 months after index PCI
  Re-hospitalization due to cardiac cause during follow-up
Cerebrovascular events | 12 months after index PCI
  ischemic or hemorrhagic stroke during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data, analytic methods, and study materials will not be made available to other researchers for purposes of reproducing the results or replicating the procedure.